CLINICAL TRIAL: NCT02093689
Title: A Phase 3 Randomized, Double-Masked, Placebo-Controlled Study of the Effect of OMS302 on Intraoperative Pupil Diameter in Subjects at High Risk of Intraoperative Floppy Iris Syndrome Undergoing Intraocular Lens Replacement Surgery
Brief Title: Intraoperative Floppy Iris Syndrome Undergoing Intraocular Lens Replacement Surgery
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Pupil measurement methodology determined not appropriate in this population.
Sponsor: Omeros Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OMS302-ILR-006
Record Dates: First submitted 2014-03-18; First posted 2014-03-21 (Estimated); Results first posted 2018-03-13 (Actual); Last update posted 2018-03-13 (Actual); Status verified 2016-11

CONDITIONS: Intraocular Lens Replacement; Intraoperative Floppy Iris Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Part 1 OMS302 (Experimental): OMS302 diluted in balanced salt solution (BSS) and administered as irrigation solution
  Interventions: Drug: Part 1 OMS302
- Part 2 OMS302 (Experimental): OMS302 diluted in balanced salt solution (BSS) and administered as irrigation solution
  Interventions: Drug: Part 2 OMS302
- Part 2 Placebo (Placebo Comparator): Placebo contains 20mM sodium citrate diluted in BSS and administered as irrigation solution.
  Interventions: Drug: Part 2 Placebo

INTERVENTIONS:
Drug: Part 1 OMS302 — OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5-mL solution containing 60.75 mM phenylephrine HCl (12.37 mg/mL) and 11.25 mM ketorolac trometamol (4.24 mg/mL) formulated in a 20 mM sodium citrate buffer (pH 6.3 ± 0.5). For administration to patients, 4.0 mL of the drug product is added to a 500-mL bottle of commercially available irrigation solution.
  Arms: Part 1 OMS302
Drug: Part 2 OMS302 — OMS302 drug product will be supplied as a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5-mL solution containing 60.75 mM phenylephrine HCl (12.37 mg/mL) and 11.25 mM ketorolac trometamol (4.24 mg/mL) formulated in a 20 mM sodium citrate buffer (pH 6.3 ± 0.5). For administration to patients, 4.0 mL of the drug product is added to a 500-mL bottle of commercially available irrigation solution.
  Arms: Part 2 OMS302
Drug: Part 2 Placebo — Placebo drug product is a sterile, clear colorless liquid, free from particulates of foreign matter. Each vial contains a nominal 4.5 mL of solution containing 20 mM sodium citrate buffer (pH 6.3 ± 0.5). For administration to patients, 4.0 mL of the drug product is added to a 500-mL bottle of commercially available irrigation solution.
  Arms: Part 2 Placebo

SUMMARY:
The purpose of this study is to evaluate the effect of OMS302 on the signs of Intraoperative Floppy Iris Syndrome in patients at risk.

DETAILED DESCRIPTION:
OMS302 is a mydriatic/anti-inflammatory combination investigational drug product being developed for use during intraoperative lens replacement (ILR). This study evaluates the effect of OMS302 on the signs of Floppy Iris Syndrome in subjects with a history of tamsulosin exposure who are undergoing ILR.

ELIGIBILITY:
Inclusion Criteria:

1. Competent to provide informed consent.
2. Voluntarily provide informed consent and HIPAA Authorization in accordance with local regulations and governing IEC/IRB requirements prior to any procedures or evaluations performed specifically for the sole purpose of the study.
3. Indicate they understand and are able, willing, and likely to fully comply with study procedures and restrictions.
4. Are male and 18 years of age or older at the time of surgery.
5. Are to undergo unilateral primary ILR, under topical anesthesia, with insertion of an intraocular lens.
6. Have a best-corrected visual acuity (BCVA) of 20/400 or better in the non-study eye.
7. Have an intraocular pressure (IOP) between 5 mm Hg and 22 mm Hg, inclusive, in the study eye.
8. Is currently and has been taking tamsulosin (Flomax®) for at least six months.

Exclusion Criteria:

1. Hypersensitivity to phenylephrine, ketoprofen, bromfenac, or other NSAIDs, including aspirin.
2. Hypersensitivity to tetracaine, lidocaine, ophthalmic viscoelastic devices (such as hydroxypropylmethylcellulose or hyaluronic acid or latex..
3. Presence of clinically significant gastrointestinal, cardiovascular, hepatic, renal, hematological, endocrine, neurological, psychiatric, respiratory or other medical condition that could increase the risk to the subject as determined by the Investigator.
4. Presence of any connective tissue disorder (e.g., lupus, rheumatoid arthritis, fibromyalgia).
5. Presence of systolic blood pressure of greater than 170 mmHg or less than 90 mmHg, or diastolic blood pressure of greater than110 mmHg or less than 40 mmHg at the screening visit.
6. Use of phenylephrine in the study eye (other than for the screening ophthalmological examination) within seven days prior to the day of surgery.
7. Use of monoamine oxidase inhibitors within 21 days prior to the day of surgery.
8. Use of pilocarpine in the study eye within seven days prior to the day of surgery.
9. Presence of narrow-angle glaucoma or unstable glaucoma.
10. Glaucoma being treated with prostaglandins or prostaglandin analogues such as Xalatan®, Lumigan®, Travatan®, and Rescula®, or Alphagan® (brimonidine tartrate) in either eye during the seven days prior to screening and through Day 7 postoperatively.
11. Presence of pseudo-capsular exfoliation in either eye.
12. History of iritis, or of any ocular trauma with iris damage in the study eye.
13. Presence of uncontrolled chronic ocular diseases in either eye that could affect pupil dilation.
14. Presence of active corneal pathology in either eye (except superficial punctate keratopathy in the non-study eye).
15. Presence of extraocular/intraocular inflammation in either eye.
16. Presence of active bacterial and/or viral infection in either eye.
17. Participating in any investigational drug or device trial within the 30 days prior to the day of surgery.
18. History of intraocular non-laser surgery in the study eye within the three months prior to the day of surgery, or intraocular laser surgery in the study eye within 30 days prior to the day of surgery.
19. Presence of any condition that the Investigator believes would put the subject at risk or confound the interpretation of the study data.
20. Investigators, employees of the investigative site, and their immediate families. Immediate family is defined as the Investigator's or employees' current spouse, parent, natural or legally adopted child (including a stepchild living in the Investigator's household), grandparent, or grandchild.
21. Prior participation in a clinical study of OMS302.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2014-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Steve Whitaker, MD, Study Director — Omeros Corporation
Locations (2):
- Omeros Investigational Site, Vienna, Austria
- Omeros Investigational Site, Bochum, Germany

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Part 2 of the study was not performed.
Groups:
- Part 2 Placebo: Placebo contains 20mM sodium citrate diluted in BSS and administered as irrigation solutions.
Period: Overall Study
Arm/Group | Part 1 OMS302 | Part 2 OMS302 | Part 2 Placebo
Started | 18 | 0 | 0
Completed | 14 | 0 | 0
Not Completed | 4 | 0 | 0
Not completed — Physician Decision | 4 | 0 | 0

BASELINE CHARACTERISTICS:
Population: All participants who had surgery were included in the analysis
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1 OMS302 | Part 2 OMS302 | Part 2 Placebo | Total
Number analyzed (Participants) | 14 | 0 | 0 | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 |  |  | 0
  Between 18 and 65 years | 0 |  |  | 0
  >=65 years | 14 |  |  | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 14 | 0 | 0 | 14

OUTCOME MEASURES:

1. Primary Outcome: Change in Pupil Diameter
Description: Change in pupil diameter over time from surgical baseline to the end of the surgical procedure determined by video capture during ILR.
Time Frame: Intraoperative
Population: Pupil measurement methodology determined not to be appropriate in this population and data were not analyzed from any participant.
Arm/Group | Part 1 OMS302 | Part 2 OMS302 | Part 2 Placebo
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: AEs are collected from time of informed consent through study completion, up to 7 days.
Arm/Group | Part 1 OMS302
Serious Adverse Events (participants affected / at risk) | 0/14
Other Adverse Events (participants affected / at risk) | 3/14
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1 OMS302 (N=14)
Zonulolysis (Eye disorders) | 1 (1)
Intraocular pressure increased (Eye disorders) | 2 (2)
Iridocele (Eye disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
This study had 2 parts. Part 1 evaluated the feasibility of the pupil measurement methodology in this patient population. The methodology was found not to be appropriate in this population. Therefore, part 2 of the study was not conducted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The data resulting from the Study was to be made public by the sponsor at the end of the study after all results were available and analyzed, with a report on the study to have been prepared in consultation with the PI, rather than being published by the PI.